CLINICAL TRIAL: NCT02840760
Title: Repetitive Transcranial Magnetic Stimulation for the Treatment of the Tardive Dyskinesia.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15ZR1435600
Record Dates: First submitted 2016-07-19; First posted 2016-07-21 (Estimated); Last update posted 2018-02-26 (Actual); Status verified 2017-06

CONDITIONS: Tardive Dyskinesia
Keywords: tardive dyskinesia.; rTMS
MeSH Terms: conditions — Tardive Dyskinesia | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- tardive dyskinesia group (Active Comparator): tardive dyskinesia group will be delivered at an intensity that is 80% of the resting motor threshold (RMT). Stimulation will be delivered at 10 Hz with 60 stimulation trains of 30 stimuli each (i.e., 1800 stimuli) and an intertrain interval of 12 sec in primary motor cortex（M1）.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation
- Healthy control group (No Intervention)

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation — Stimulate the primary motor cortex for 2 weeks.
  Arms: tardive dyskinesia group

SUMMARY:
The purpose of this study is to explore the therapeutic effect and mechanism of transcranial magnetic stimulation (rTMS) in the treatment of the tardive dyskinesia.

DETAILED DESCRIPTION:
The study was a parallel control design trial for 2 weeks. Patients with schizophrenia were treated with 10-Hz rTMS on left motor cortex (added to the ongoing treatment). Clinical symptoms and MEP were assessment before and after rTMS treatment.

ELIGIBILITY:
Inclusion Criteria:

* The diagnosis of schizophrenia according to DSM-IV；
* At least two item of Abnormal Involuntary Movement Scale（AIMS） must be 2 points or higher
* these symptoms are not from Parkinson，tourette's syndrome,huntington disease
* Signed an informed consent

Exclusion Criteria:

* rTMS contraindications: intracranial metal substance, with heart pacemakers and cochlear implants, intracranial pressure
* patients to be diagnosed according to DSM-IV for substance abused, development delayed
* current treatment with anticonvulsant acting drugs such as anticonvulsants, benzodiazepines
* Acute risk of suicide and impulse
* history of epileptic seizures or the presence of epileptic activity documented on the basis of EEG
* pregnant and lactant women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-09 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in motor evoked potential(MEP) | 2 times (Before treatment,immediately after treatment)
Change from baseline in Abnormal Involuntary Movement Scale(AIMS） | 2 times (Before treatment,immediately after treatment)

SECONDARY OUTCOMES:
Change from baseline in cortical silent period | 2 times (Before treatment,immediately after treatment)
Change from baseline in short interval intracortical inhibition(SICI） | 2 times (Before treatment,immediately after treatment)
Change from baseline in intracortical facilitation(ICF） | 2 times (Before treatment,immediately after treatment)
Change from baseline in Simpson-Angus Scale（SAS） | 2 times (Before treatment,immediately after treatment)
Change from baseline in Barnes Akathisia Rating Scale（BARS） | 2 times (Before treatment,immediately after treatment)
Change from baseline in Positive and Negative Syndrome Scale（PANSS） | 2 times (Before treatment,immediately after treatment)
Change from baseline in clinical global impression (CGI) | 2 times (Before treatment,immediately after treatment)

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Mental Health Center, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No